CLINICAL TRIAL: NCT00832585
Title: A Phase IV, Open Label Study to Evaluate the Safety and Efficacy of Intramuscular (IM) Alefacept (Amevive) 15mg/wk in Subjects 18 Years and Older With Moderate to Severe Atopic Dermatitis
Brief Title: Study to Evaluate the Safety and Efficacy of Alefacept (Amevive) in Subjects With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Michael D. Tharp, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC 07-001
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Results first posted 2011-01-28 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic; Dermatitis; chronic; skin
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Bronchiolitis Obliterans Syndrome | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alefacept (Experimental): Amevive® has been shown to be a safe and effective agent in the treatment of psoriasis but may prove useful in treating atopic dermatitis at a dose of 15mg IM every week for 12 weeks. Unlike other "biologics" for the treatment of skin diseases, the use of alefacept is not associated with increased infection, congestive heart failure, demyelinating disorders or lupus- like syndromes.
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — Alefacept 15mg IM every week for 12 weeks
  Other Names: Amevive

SUMMARY:
This study will assess the safety, tolerability, and efficacy of Alefacept in patient with moderate to severe atopic dermatitis who could not be adequately controlled with topical therapies.

DETAILED DESCRIPTION:
Atopic dermatitis is a chronic inflammatory skin disease associated with cutaneous hyper-reactivity to environmental triggers that are generally innocuous to healthy, nonatopic individuals (Leung et al. 2004). Acute eczematous skin lesions in atopic dermatitis are characterized by marked epidermal intercellular edema (spongiosis). Chronic lesions are characterized by an acanthotic epidermis with elongation of the rete ridges, parakeratosis, and minimal spongiosis (Leung and Bieber 2003).

A significant mixed inflammatory cell infiltrate is present in both acute and chronic skin lesions, consisting of lymphocytes, immunoglobulin E (IgE)-bearing Langerhans cells, inflammatory dendritic epidermal cells, and macrophages. Eosinophils are also present in varying levels (Leung and Bieber 2003).

Activation and skin-selective homing of peripheral blood T lymphocytes and their subsequent effector functions in the skin represent sequential immunologic events in the pathogenesis of atopic dermatitis (Akdis et al. 2000). More than 90% of skin-infiltrating T lymphocytes in inflammatory skin diseases such as atopic dermatitis express CD44- and the oligosaccharide determinant cutaneous lymphocyte-associated antigen (CLA) (Berg et al. 1991). The migration of CD4+, CLA-positive T lymphocytes across cytokine-activated endothelial cell layers has 2 been shown to be dependent on the interaction of lymphocyte function-associated antigen (LFA)-1 and intercellular adhesion molecule (ICAM)-1 (Santamaria Babi et al. 1995).

The activation of T lymphocytes plays an important role in atopic dermatitis pathogenesis. In acute atopic dermatitis, a T-helper (TH)2 cytokine profile is predominantly seen, with increased expression of interleukin (IL)-4, lL-5, and IL-13 (Stone 2003). In chronic atopic dermatitis, the cytokine profile changes to a TH1 predominant profile, with increased expression of interferon y (IFN-y) (Leung et al. 2004). Activated T lymphocytes also are responsible for direct cell-mediated keratinocyte apoptosis, which contributes to the spongiosis pattern of epidermal injury characteristic of acute atopic dermatitis (Trautmann et al. 2001),

The interaction of T lymphocytes with antigen-presenting cells (APCs) is one of the initial steps in T lymphocyte activation of an immunologic response to what is perceived by the immune system to be a foreign antigen. Although much attention has been focused on the primary interaction of the T lymphocyte receptor with the major histocompatability complex (MHC)-antigen complex on the APC, several other cell surface components are also involved in, and necessary for, T lymphocyte activation. Ligand pairs necessary for T lymphocyte activation, located on the cell surface of the T lymphocytes and the APC, respectively, include CD2/LFA-3, LFA-1/ICAM-1 (also ICAM-2 and ICAM-3), CD281B7, CD4/MHC Class II, and CD8/MHC Class I. CD2 interaction with LFA.-3 is necessary for T lymphocyte activation, binding, and T-helper cell responses. (Fischer et al. 1986; Springer et al. 1987)

Anievive® (Alefacept) is a dimeric fusion protein that consists of the extracellular CD2 binding portion of the human leukocyte function antigen -3 (LFA-3) linked to the Fc portion of IgG1. Amevive® interferes with lymphocyte activation by specifically binding to CD2 on lymphocytes thereby inhibiting LFA-3/CD2 interaction. Amevive® causes a reduction in CD4+ lymphocytes which play a role in atopic dermatitis. Currently, Amevive® has been shown to be a safe and effective agent in the treatment of psoriasis but may prove useful in treating atopic dermatitis. Unlike other "biologics" for the treatment of skin diseases, the use of alefacept is not associated with increased infection, congestive heart failure, demyelinating disorders or lupus- like syndromes. (1-Lodak and David, 2004)

Ten atopic patients who meet the inclusion/exclusion criteria will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form(s)
* Age of l8 years or older
* A diagnosis of atopic dermatitis as determined by the diagnostic criteria for atopic dermatitis
* Disease severity of 3 or 4 (moderate or severe) as assessed by PGA rating (0-4 scale)
* Be a candidate for systemic therapy who cannot be adequately controlled (ie have a PGA assessment of 3 014) with topical therapies (Le., medium-to high-potency topical corticosteroids, tacrolimus, or pimecrolimus).
* For female subjects of childbearing potential, use of an acceptable method of contraception to prevent pregnancy and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study and for 3 months after the last dose of Alefacept
* Willingness to hold sun exposure reasonably constant and to avoid use of tanning booths or other ultraviolet (UV) light sources during the study

Exclusion Criteria

* History of hypersensitivity to alefacept or any of its components
* History of illegal drug or alcohol abuse
* History of or ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
* History of eczema herpeticum within the 30 days prior to screening
* History of opportunistic infections (e.g., systemic fungal infections, parasites)
* History of hepatitis B or C virus
* History of active tuberculosis (TB) or currently undergoing treatment for TB.
* Presence of history of malignancy within the past 5 years, including lymphoproliferative disorders. Subjects with a history of fully resolved basal cell or squamous cell skin cancer may be enrolled in the study
* Pregnant or lactating women
* Diagnosis of hepatic cirrhosis, regardless of cause or severity
* Hospital admission for cardiovascular or pulmonary disease within the year prior to screening, including hospitalization for asthma exacerbations
* Subjects admitted to the hospital for chest pain that was subsequently determined to be non-cardiac in origin may be enrolled
* History of clinically significant anemia
* WBC count <4000/pL or> 14,000/pL
* Use of experimental drugs or treatments within 30 days or 5 half-lives, whichever is longer, prior to the first dose of alefacept
* Use of a live virus or live bacteria vaccine in the 14 days prior to be the first dose of alefacept
* Any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to study drug or would significantly interfere with the subject's ability to comply with the provisions of this protocol
* Any subject whose baseline atopic dermatitis PGA rating has changed to 0, 1, or 2 (clear, almost clear, or mild) from a screening rating of 3,4, or 5 (moderate, severe, or very severe)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Tharp, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center - Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from physician referrals and advertisements placed within the Rush University Medical Center campus. Recruitment was opened between Jan 08 through Sept 09
Groups:
- Alefacept: Amevive® has been shown to be a safe and effective agent in the treatment of psoriasis but may prove useful in treating atopic dermatitis. Unlike other "biologics" for the treatment of skin diseases, the use of alefacept is not associated with increased infection, congestive heart failure, demyelinating disorders or lupus- like syndromes. The dose for Alefacept is 15mg, the dosage form is intramuscular injection (IM), and the frequency of administration is once a week for 12 weeks.
Period: Overall Study
Arm/Group | Alefacept
Started | 5 (Eight subjects were screened but only 5 started the study and received study drug.)
Completed | 3 (Only three subjects completed all of the visits for the study as per protocol.)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alefacept
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.84 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Eczema Area Severity Index (EASI) Score From Baseline (Week 1) to Week 16.
Description: The Eczema Area Severity Index (EASI) measures erythema (E), infiltration (I), excoriation (Ex) and lichenification (L) using 0=none, 1=mild, 2=moderate, 3=severe. Head/neck, upper limbs, trunk, lower limbs are rated from 1 to 6 (0=no eruption, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89%, 6=90-100%). The proportional factor for the head/neck =.01, upper limbs=.02, trunk=.03 and lower limbs=.04. The algorithm for calculating the EASI is the sum of E+I+Ex+L multiplied by the area, multiplied by the proportional factor. The total score is the sum of the four body-region scores, max=72, min=0.
Time Frame: Week 1 to week 16
Population: 8 (4 female and 4 male) atopic patients, ranging in age from 24 to 54 yrs of age, were screened for the study. 5 patients were enrolled for 12 wks of treatment, but only 3 completed the study.
Measure: Median (Full Range); unit: Scores on a scale.
Arm/Group | Alefacept
Number analyzed (Participants) | 3
Scores on a scale. | 26.4 [13.2 to 29.8]

2. Secondary Outcome: Change in Physician Global Assessment (PGA) Score From Baseline (Week 1) to Week 16.
Description: The Physician Global Assessment (PGA) evaluates the overall severity of Atopic Dermatitis (AD) at a given time using a four point scale (0=clear, 0.5=clear to mild, 1=mild, 1.5=mild to moderate, 2=moderate, 2.5=moderate to severe, and 3=severe).
Time Frame: Week 1 to week 16
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Alefacept
Number analyzed (Participants) | 3
Scores on a scale | 1 [1 to 1.5]

ADVERSE EVENTS:
Arm/Group | Alefacept
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alefacept (N=5)
Joint Infection (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No